CLINICAL TRIAL: NCT06269172
Title: PAINT Breathlessness
Brief Title: Perceptions Across Ethnicities to Develop an Adapted Intervention for Breathlessness
Acronym: Paint
Status: Recruiting | Type: Observational
Sponsor: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 162076; 322453 (Other: HRA)
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: intereviews — An individual's experience of their breathlessness is influenced by multiple factors including their medical condition, psychology, sociological and situational circumstances which will include ethnicity. There is currently a lack of evidence exploring the impact of ethnicity in the experience and presentation of breathlessness.
  The non-medical management of breathlessness in respiratory diseases includes pulmonary rehabilitation (PR). PR is a highly evidenced exercise-based intervention to help manage breathlessness, improving health-related quality of life and improving survival. Recent audits in England and Wales showed 89% of patients attending PR were recorded as having a White British ethnicity which is in contrast to national ethnicity demographics. This may be because the cultural acceptability of PR components are not fully considered.

SUMMARY:
An individual's experience of their breathlessness is influenced by multiple factors including their medical condition, psychology, sociological and situational circumstances which will include ethnicity. There is currently a lack of evidence exploring the impact of ethnicity in the experience and presentation of breathlessness.

The non-medical management of breathlessness in respiratory diseases includes pulmonary rehabilitation (PR). PR is a highly evidenced exercise-based intervention to help manage breathlessness, improving health-related quality of life and improving survival. Recent audits in England and Wales showed 89% of patients attending PR were recorded as having a White British ethnicity which is in contrast to national ethnicity demographics. This may be because the cultural acceptability of PR components are not fully considered. Therefore, this study will explore how individuals with cardiorespiratory disease from different ethnicities from the Leicestershire population experience and manage their breathlessness through art workshops, focus groups and interviews. Informed by these results, the study team will work with individuals from under-represented ethnicities and key stakeholders to co-design adaptations of PR that may improve the management of breathlessness in underrepresented ethnicities that do not attend conventional PR programmes.

The study is funded by the Wellcome Trust as part of the Leicestershire Health Inequalities Improvement Programme at the University of Leiceste

DETAILED DESCRIPTION:
An individual's experience of their breathlessness is influenced by multiple factors including their medical condition, psychology, sociological and situational circumstances which will include ethnicity. There is currently a lack of evidence exploring the impact of ethnicity in the experience and presentation of breathlessness.

The non-medical management of breathlessness in respiratory diseases includes pulmonary rehabilitation (PR). PR is a highly evidenced exercise-based intervention to help manage breathlessness, improving health-related quality of life and improving survival. Recent audits in England and Wales showed 89% of patients attending PR were recorded as having a White British ethnicity which is in contrast to national ethnicity demographics. This may be because the cultural acceptability of PR components are not fully considered. Therefore, this study will explore how individuals with cardiorespiratory disease from different ethnicities from the Leicestershire population experience and manage their breathlessness through art workshops, focus groups and interviews. Informed by these results, the study team will work with individuals from under-represented ethnicities and key stakeholders to co-design adaptations of PR that may improve the management of breathlessness in underrepresented ethnicities that do not attend conventional PR programmes.

The study is funded by the Wellcome Trust as part of the Leicestershire Health Inequalities Improvement Programme at the University of Leiceste

ELIGIBILITY:
Inclusion Criteria:

* Stage 1: Art Workshops, Focus Groups and Semi-Structured Qualitative Interviews Willing and able to provide informed consent for participation in the art workshop, focus group/semi-structured qualitative interview Any individual over 18 years across ethnicities Able to communicate in spoken and written English OR Art workshop and interview: translator for an individuals preferred spoken and written language is available.

Identifies as Grades 2-5 on the Medical Research Council Dyspnoea Scale (MRC). Eligible for PR (e.g., confirmed respiratory condition, functional limitations due to breathlessness).

Stage 2: Experience Based Co-design Willing and able to provide informed consent for participation in the co-design process.

Any individual over 18 years Able to communicate in spoken and written English or a translator for their spoken and written language is available.

Eligible for PR (e.g., confirmed respiratory condition, functional limitations due to breathlessness) and identifies as an ethnicity that the intervention is being adapted for or a family member, friend or carer of an individual with breathlessness that is eligible for PR and identifies as an ethnicity that the intervention is being adapted for OR works for healthcare provider in a service that refers to or delivers PR OR is a charity representative.

Able to attend co-design workshops

Exclusion Criteria:

* Stage 1: Art Workshop, Focus Groups and Semi-Structured Qualitative Interviews Unable to provide informed consent Any individual under 18 years Art workshop and interview: If no translator available. Focus group only: not able to speak English due to group interaction required. Identifies as Grade 1 on the MRC scale. Not eligible for PR (e.g. any significant comorbidities which limits exercise training ability).

Stage 2: Experience Based Co-design Unable to provide informed consent. Any individual under 18 years If no translator is available. Not eligible for PR or does not identify as an ethnicity that the intervention is being adapted for OR a family member, friend or client is not eligible for PR or does not identify as an ethnicity that the intervention is being adapted for OR does not work for a healthcare provider in a service that refers to or delivers PR OR is not a charity representative.

Unable to attend co-design workshops

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: cardiovascular
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Art Workshops, Focus Groups and Semi-Structured Interviews | 21 months
  stage 1

SECONDARY OUTCOMES:
: Experience Based Co-design The co-development of an intervention for breathlessness for under-represented ethnicities. | 21 months
  Stage 2

CONTACTS AND LOCATIONS:
Locations (1):
- Glenfield Hospital, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No